CLINICAL TRIAL: NCT03280407
Title: NEOadjuvant Chemotherapy Only Compared With Standard Treatment for Locally Advanced Rectal Cancer: a Randomized Phase II Trial
Brief Title: NEOadjuvant Chemotherapy Only Compared With Standard Treatment for Locally Advanced Rectal Cancer
Acronym: NEOLAR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Ismail Gögenur, Professor, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-20160158
Record Dates: First submitted 2017-09-07; First posted 2017-09-12 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Colorectal Neoplasm; Colorectal Cancer; Rectal Neoplasms; Chemotherapy Effect; Intestinal Disease; Intestinal Neoplasms; Rectal Cancer
Keywords: Neoadjuvant chemotherapy,; locally advanced rectal cancer,; chemotherapy; CAPOX (oxaliplatin/capecitabine); FOLFOX (oxaliplatin/leucovorin/5FU)
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms; Intestinal Diseases; Intestinal Neoplasms | interventions — Capecitabine; Folfox protocol; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: This is an open label, randomized phase II screening trial allocating eligible patients to either standard treatment for rectal cancer or experimental preoperative combination chemotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A, capecitabine (Active Comparator): Radiochemotherapy with 50.4 Gy in 28 fractions concomitantly with chemotherapy
  Interventions: Drug: Capecitabine
- B, FOLFOX or CAPOX (Experimental): Neoadjuvant chemotherapy with CAPOX (oxaliplatin/capecitabine) or FOLFOX regimen (oxaliplatin/leucovorin/5FU), according to institutional practice
  Interventions: Drug: FOLFOX regimen (oxaliplatin/leucovorin/5FU); Drug: CAPOX (oxaliplatin/capecitabine)

INTERVENTIONS:
Drug: Capecitabine — Radio-chemotherapy with 50.4 Gy in 28 fractions to tumor and regional lymph nodes concomitantly with capecitabine 825 mg/m2 b.i.d
  Arms: A, capecitabine
Drug: FOLFOX regimen (oxaliplatin/leucovorin/5FU) — Six cycles: Oxaliplatin 85 mg/m2 day 1, leucovorin 400 mg/m2 day 1, 5FU 400 mg/m2 bolus day 1 and 5FU 2400 mg/ m2 over 46-48 hours day 1-3, repeated every two weeks.
  Other Names: FOLFOX (oxaliplatin/leucovorin/5FU)
  Arms: B, FOLFOX or CAPOX
Drug: CAPOX (oxaliplatin/capecitabine) — Four cycles: Oxaliplatin 130 mg/m2 day 1 and capecitabine 1000 mg/m2 b.i.d. days 1-14, repeated every 3 weeks.
  Arms: B, FOLFOX or CAPOX

SUMMARY:
The main clinical hypothesis is that compared to radio-chemotherapy for low and mid rectal tumors or surgery for high rectal tumors neoadjuvant chemotherapy reduces the rate of distant relapse without increasing the rate of local relapse.

The aim of the present study is to compare long term and short term outcomes in rectal cancer patients undergoing standard treatment (radio-chemotherapy/surgery) or experimental neoadjuvant chemotherapy/surgery Furthermore, early surgical and medical complications, the functional outcome, toxicity and quality of life (QoL) may be improved if radiotherapy can be avoided.

Exploratory analyses are planned in order to find potential predictive markers for selecting patients to either radio-chemotherapy/surgery or neoadjuvant combination chemotherapy/surgery.

DETAILED DESCRIPTION:
The standard treatment of locally advanced but resectable cancer in the middle or lower rectum is preoperative radio-chemotherapy and in the upper part initial surgery. The clinical benefit from radio-chemotherapy is primarily through a reduction in local relapse but the treatment is associated with acute toxicity and long term functional dysfunction. Subsequently, it is important to select patients with high risk of local relapse. Intense systemic combination chemotherapy reduces the risk of distant relapse and increases survival in the postoperative setting. The biological rationale is eradication of micrometastases and hence it may be anticipated that earlier, i.e. neoadjuvant, combination therapy may improve systemic control.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the rectum with the lower boarder within 15 cm from the anal verge
* Locally advanced tumor based on imaging
* T3 tumors within 10 cm from the anal verge fulfilling the criteria for preoperative radio-chemotherapy according to Danish Colorectal Cancer Group (DCCG) guidelines
* T3c or T4 tumors 10-15 cm from the anal verge
* Deemed resectable at the multidisciplinary team (MDT) conference
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Age at least 18 years
* Adequate bone marrow, liver and renal function allowing systemic chemotherapy
* Absolute neutrophil count ≥1.5x109/l and thrombocytes ≥ 100x109/l.
* Bilirubin ≤ 1.5 x upper normal value and alanine aminotransferase ≤ 3 x upper normal value
* Calculated or measured renal glomerular filtration rate at least 30 mL/min
* Anticonception for fertile women and for male patients with a fertile partner. Intrauterine device, vasectomy of a female subject's male partner or hormonal contraceptive are acceptable
* Written and orally informed consent

Exclusion Criteria:

* Distant metastasis
* Invasive ingrowth into other organs
* Incapacity, frailty, disability and comorbidity to a degree that according to the investigator is not compatible with combination chemotherapy
* Previous radiotherapy to the pelvis
* Previous treatment with 5FU or oxaliplatin
* Surgery within two weeks
* Neuropathy NCI grade > 1
* Other malignant tumor within 5 years except non-melanoma skin cancer or carcinoma in situ cervicis uteri
* Pregnant (positive pregnancy test) or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 5 years
  All patients will be evaluated with CT and MRI scans and clinically every 6 months for 2 years and annually until the number of events is reached and the trial is stopped (max 5 years)

SECONDARY OUTCOMES:
Overall survival | 5 years
  All patients will be evaluated with CT and MRI scans and clinically every 6 months for 2 years and annually for maximum 5 years
Local relapse | 5 years
  Defined to be within the pelvis. Any relapse should be verified by biopsy
Distant relapse | 5 years
  Defined to be outside the pelvis. Any relapse should be verified by biopsy
Early toxicity | 5 years
  Evaluated using CTCEA (Common Terminology Criteria for Adverse Events) version 4.
Late toxicity | 5 years
  Evaluated using CTCEA version 4.
Functional outcome | 5 years
  Measured with LARS questionnaire
Quality of life (QoL) | 5 years
  Measured with EORTC QoL questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Gögenur, MD, Study Chair — Department of Surgery, ZUH; Lars Henrik Jensen, MD, Principal Investigator — Vejle Hospital
Locations (1):
- Vejle Hospital, Vejle, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Undecided